CLINICAL TRIAL: NCT07008599
Title: Assessment of Inflammatory Biomarkers in Molar-Incisor Hypomineralization-Affected First Permanent Molars: A Controlled Clinical Study
Brief Title: Assessment of Inflammatory Biomarkers in Molar-Incisor Hypomineralization-Affected First Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Seray Şahin, Principal Investigator, Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MUPEDODENTSERAYSAHİN
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-05

CONDITIONS: Molar-Incisor Hypomineralization (MIH); Pulp Disease, Dental; Inflamation
Keywords: Molar-Incisor Hypomineralization (MIH); Tooth Hypersensitivity; Pediatric Dentistry; Pulpal Biomarkers
MeSH Terms: conditions — Molar Hypomineralization; Dental Pulp Diseases; Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MIH Asymptomatic (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample
- MIH Reversible (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample
- MIH Irreversible (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample
- Control Asymptomatic (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample
- Control Reversible (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample
- Control Irreversible (Other): Pulp blood samples were collected during the procedure of vital pulp treatment
  Interventions: Other: Pulpal Blood Sample

INTERVENTIONS:
Other: Pulpal Blood Sample — Biochemical markers were measured in blood samples using enzyme-linked immunosorbent assay (ELISA).

SUMMARY:
Molar-Incisor Hypomineralization (MIH) is a qualitative developmental defect of enamel primarily affecting the permanent first molars and often incisors. The global prevalence of MIH ranges from 2.9% to 44%. Although the precise etiology of MIH remains unclear, it is considered multifactorial, involving interactions between genetic, environmental, and systemic factors during the prenatal, perinatal, and postnatal periods. Environmental toxins such as Bisphenol A (BPA) have also been implicated in its development. Despite the well-documented impact of MIH on enamel and dentin, little is known about the inflammatory changes in the pulp tissue of these teeth. This controlled clinical study aims to assess the levels of proinflammatory and anti-inflammatory cytokines in the pulp tissues of first permanent molars affected by MIH and compare them with those in non-MIH teeth. The null hypothesis is that there is no statistically significant difference in the levels of these cytokines between MIH-affected and non-affected pulp tissues. The findings are expected to contribute valuable insights into the pathophysiology of MIH-related pulpal involvement and support the development of improved diagnostic and therapeutic strategies. Pulpal blood samples were obtained from 85 first permanent molars of systemically healthy children aged 8 to 13 who underwent pulp therapy. Based on the presence or absence of Molar-Incisor Hypomineralization (MIH), teeth were assigned to either the MIH group or the control group. To evaluate the dental status and detect possible signs of pulpitis, the MIH-TNI index, Schiff sensitivity scale, Periapical Index (PAI), cold test responses, and other clinical parameters were recorded.

DETAILED DESCRIPTION:
Molar-Incisor Hypomineralization (MIH) is a qualitative developmental enamel defect that predominantly affects the permanent first molars and frequently involves incisors. Characterized by demarcated opacities and structurally compromised enamel, MIH increases the susceptibility of teeth to post-eruptive breakdown, rapid caries progression, and functional and aesthetic impairments. Globally, MIH prevalence ranges from 2.9% to 44%, and in Turkey, it has been reported between 7.7% and 24%, indicating significant public health relevance.

The etiology of MIH is considered multifactorial, involving complex interactions among genetic, systemic, and environmental factors across prenatal, perinatal, and postnatal periods. Environmental toxins, such as bisphenol A (BPA), and systemic conditions like low birth weight, preterm birth, and early childhood illnesses, have been implicated. Microscopic studies demonstrate decreased mineral content, altered hydroxyapatite crystal structure, and reduced microhardness in MIH-affected enamel. These properties compromise enamel integrity, facilitate bacterial penetration, and increase the risk of pulpal involvement. MIH-affected dentin typically exhibits widened dentinal tubules, increasing dentin permeability and promoting rapid stimulus transmission to the pulp. Clinically, this is associated with hypersensitivity, difficulty in achieving anesthesia, and pulpal inflammation. However, the specific inflammatory profiles of pulps in MIH-affected teeth have not been thoroughly studied.

This controlled clinical study aims to investigate and compare the levels of proinflammatory (TNF-α, IL-6, IL-8) and anti-inflammatory (IL-4, IL-10, IL-13) cytokines, as well as tissue degradation markers (MMP-3, MMP-8, MMP-9), in the pulpal blood of MIH-affected versus non-affected first permanent molars.

A total of 85 first permanent molars requiring pulp therapy were selected from systemically healthy children aged 8 to 13 years. Based on MIH status, the teeth were categorized into MIH and control groups. Clinical evaluation included assessment using the MIH Treatment Need Index (MIH-TNI), Schiff Cold Air Sensitivity Scale, Periapical Index (PAI), cold test responses, and other clinical signs of pulpitis. Pulpal blood samples were collected under sterile conditions using cotton pellets, transferred into lithium heparin-coated tubes, and stored at -70°C. Enzyme-linked immunosorbent assay (ELISA) was used to quantify the levels of TNF-α, IL-4, IL-6, IL-8, IL-10, IL-13, MMP-3, MMP-8, and MMP-9. This study is expected to provide novel insights into the pathophysiology of MIH-related pulp inflammation and contribute to the development of improved diagnostic and treatment strategies in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 13 years who were cooperative (able to comply with instructions)
* Without any systemic diseases, syndromes, anomalies, or known allergies
* First permanent molars requiring pulp therapy were included in the study.

Exclusion Criteria:

* Patients who had used antibiotics within the last month
* Teeth deemed unrestorable
* Teeth showing lamina dura loss or pathological root resorption on radiographic examination
* Teeth that had previously undergone endodontic treatment
* Teeth with internal or external root resorption
* Teeth presenting with pus, necrosis, or exudate at the exposure site during treatment
* Teeth in which no pulp exposure occurred during the procedure

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of biochemical mediators in pulpal blood samples using enzyme-linked immunosorbent assay (ELISA) | 26.11.2024- 16.04.2025
  Quantitative concentrations (pg/mL) of proinflammatory (TNF-α, IL-6, IL-8) and anti-inflammatory (IL-4, IL-10, IL-13) cytokines, as well as matrix metalloproteinases (MMP-3, MMP-8, MMP-9), measured using ELISA in pulpal blood.

CONTACTS AND LOCATIONS:
Overall Officials: Seray Şahin, Doctor of Dental Surgery (DDS), Principal Investigator — Marmara University, School of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Marmara Üniversitesi Recep Tayyip Erdoğan Külliyesi Sağlık Yerleşkesi, Diş Hekimliği Fakültesi, Başıbüyük Yolu 9/3 34854 Başıbüyük / Maltepe / İSTANBUL, Istanbul, Beypazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including intraoral photographs and clinical evaluation scores) may be shared in scientific publications or presentations. Data will be limited to information relevant for scientific analysis and will not include any personal identifiers.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD), along with supporting documents such as the study protocol and statistical analysis plan, will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following the publication date.
Access Criteria: Requests for access to de-identified individual participant data and supporting documents will be considered for academic or scientific research purposes. Interested researchers must submit a written proposal detailing the planned analysis, including objectives and statistical methods. Requests will be reviewed by the principal investigator and institutional review board (IRB) representatives to ensure ethical compliance and scientific merit. A data use agreement must be signed prior to data release. Requests can be submitted via email to the corresponding author listed in the publication.